CLINICAL TRIAL: NCT05049174
Title: Clinical and Health-economic Effects of a Nurse-led Smoking Cessation Program With Follow-up in Healthy Life Centres With Free Cessation Drugs: a Randomized Clinical Trial
Brief Title: Nurse-led Smoking Cessation Program With Follow-up in Healthy Life Centres: a Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: University of Oslo (Other); Oslo University Hospital (Other); Norwegian Directorate of Health (Other Government); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 270267
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation; Smoking Behaviors; Nurse's Role; Cardiovascular Diseases
MeSH Terms: conditions — Smoking Cessation; Smoking; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1 to an in-hospital nurse-led smoking cessation intervention with systematic referrral to the municipal healthy life-centres or to written information about smoking cessation and the municipal health service program.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive intervention (Experimental)
  Interventions: Behavioral: Nuse-led interview and referral to municipal healthy life-centres
- Low-threshold intervention (Active Comparator)
  Interventions: Behavioral: Nuse-led interview and referral to municipal healthy life-centres

INTERVENTIONS:
Behavioral: Nuse-led interview and referral to municipal healthy life-centres — Usual care treatment and written information to patients and general practitionnaires about smoking cessation and the municipal healthy life-centres

SUMMARY:
A better understanding of how to incorporate effective smoking cessation measures into clinical practice is requested. In this is prospective, multi-center, randomized, open, blinded end-point (PROBE) trial, we assigned daily smokers hospitalized with an acute cardiac event 1:1 to an in-hospital nurse-led smoking cessation intervention with direct referral to further follow-up in the municipal healthy life-centres (intensive intervention) or to written information about smoking cessation and the municipal program (low-threshold intervention) . The primary outcome will be the smoking cessation rates between the groups at 6 months follow-up. Key secondary outcomes include a cost-effectiveness analysis of the intensive intervention and cessation rates at 3- and 12-months follow-up, the proportion who used nicotine replacement therapy and the proportion who attended the healthy-life center program between the two groups. We also assess effects of recurrent cardiovascular events and mortality after 12 months, two and five years follow-up. Exploratory analyses include new knowledge about the patient and system factors of importance for participation to healthy life-centers and for changes in smoking behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years and smokes at least 1 cigarette daily
* Hospitalized with an acute cardiovascular event (i.e. myocardial infarction, unstable or stable angina, arrythmias, stroke, transitory ischemic attac, carotid stenosis or claudication with need for revascularization)
* established atheroscledrotic cardiovascular disease
* Sign informed consent and is expected to participate according to ICH /GCP

Exclusion Criteria:

* Does not usually live or work in the Vestre Viken catchment area
* Any condition (e.g. psychosis, alcohol abuse, dementia) or situation that may pose a significant risk to the participant, confuse the results or make participation unethical
* Lack of Norwegian and English knowledge
* Short life expectancy (<12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference between the groups in point prevalence of self-report smoking abstinence at six months follow-up | Six months after randomization
  Difference between the groups in the proportion of participants who self-report smoking abstinence over the whole follow-up period at six months follow-up allowing up to five cigarettes in total

SECONDARY OUTCOMES:
Difference between the groups in proportion who quit smoking determined with objectively | Six months after randomization
  Difference between the groups in proportion of participants who quit smoking measured by the level of carbon monoxide in the exhaled air
Difference between the groups in point prevalence of self-report smoking abstinence three months after randomization | Three months after randomization
  Difference between the groups in the proportion of participants who self-report smoking abstinence over the whole periode follow-up period at six months follow-up allowing up to five cigarettes in total
Difference between the groups in point prevalence of self-report smoking abstinence 12 months after randomization | Twelve months after randomization
  Difference between the groups in the proportion of participants who self-report smoking abstinence over the whole periode follow-up period at six months follow-up allowing up to five cigarettes in total
Differences in participation rate at healthy life-centres between the groups | 8 to 12 weeks after randomization
  Differences in participation rate at healthy life-centres between the groups measured by telephone interview with personnell at the healthy life-centres
Differences in use of smoking cessation aids between the groups | 8 to 12 weeks after randomization
  Differences in the proportion of patients who use of smoking cessation aids (nicotine replacement therapy) between the groups measured by patient self-report
Difference between the groups in the composite end-point all-cause mortality, hospitalisation for myocardial infarction, stroke, transitrory ischemic attac, coronary revascularisation or symptomatic periperial artery disease | From baseline until 2 years follow-up
  Difference between the groups in the composite end-point all-cause mortality, hospitalisation for myocardial infarction, stroke, transitrory ischemic attac, coronary revascularisation or symptomatic periperial artery disease obtained from hospital medical records
Difference between the groups in the composite end-point all-cause mortality, hospitalisation for myocardial infarction, stroke, transitrory ischemic attac, coronary revascularisation or symptomatic periperial artery disease | From baseline until 5 years follow-up
  Difference between the groups in the composite end-point all-cause mortality, hospitalisation for myocardial infarction, stroke, transitrory ischemic attac, coronary revascularisation or symptomatic periperial artery disease obtained from hospital medical records

OTHER OUTCOMES:
Differences in changes in clinical and psychological factors between the study groups | From baseline until 6 months follow-up
  Differences between the study groups in the proportion of participants who report significant changes in clinical and psychological factors from baseline until six months follow-up measured by patient self-report

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Drammen Hospital, Drammen, Akershus
  - Ringerike Hospital, Hønefoss, Akershus
  - Kongsberg Hospital, Kongsberg, Akershus

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT05049174/SAP_001.pdf